CLINICAL TRIAL: NCT04976582
Title: Effect of the Dry Needling and Kinesio Taping in Management of Mechanical Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Responsible Party: Principal Investigator, Dr.Adeela Asad, PRINICIPAL INVESTIGATOR, Shaheed Zulfiqar Ali Bhutto Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: not applicale
Record Dates: First submitted 2020-11-11; First posted 2021-07-26 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Mechanical Low Back Pain
Keywords: kinesio-taping, dry needling, low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Participants will be divided into two groups Group 1: control group in which kinesiotaping with conventional physical therapy treatment (modalities including transcutaneous electrical nerve stimulation (TENS); electrical muscle stimulation (EMS); and interferential current (IFC). Physical agents including ultrasound, hot packs, and cold packs. Exercise including McKenzie exercises) will be administered.
  Group 2: experimental group in which dry needling with conventional physical therapy treatment modalities including transcutaneous electrical nerve stimulation (TENS); electrical muscle stimulation (EMS); and interferential current (IFC). Physical agents including ultrasound, hot packs, and cold packs. Exercise including McKenzie exercises) will be administered.
Masking Description: Researcher and participants both are familiar with the procedure of interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional group (Experimental): experimental group in which dry needling with conventional physical therapy treatment modalities including transcutaneous electrical nerve stimulation (TENS); electrical muscle stimulation (EMS); and interferential current (IFC). Physical agents including ultrasound, hot packs, and cold packs. Exercise including McKenzie exercises) will be administered.
  Interventions: Device: dry needle
- control group (No Intervention): control group in which kinesiotaping with conventional physical therapy treatment (modalities including transcutaneous electrical nerve stimulation (TENS); electrical muscle stimulation (EMS); and interferential current (IFC). Physical agents including ultrasound, hot packs, and cold packs. Exercise including McKenzie exercises) will be administered.

INTERVENTIONS:
Device: dry needle — modalities including transcutaneous electrical nerve stimulation (TENS); electrical muscle stimulation (EMS); and interferential current (IFC). Physical agents including ultrasound, hot packs, and cold packs. Exercise including McKenzie exercises) will be administered.
  Other Names: Exercise including McKenzie exercises
  Arms: interventional group

SUMMARY:
Low back pain (LBP) is an extremely common problem that most people experience at some point in their life. It is the leading cause of activity limitation and work absence throughout much of the world. In India, occurrence of LBP is also alarming. Nearly 60% of the population has significant back pain at some time in their life. In Brazil, spinal pain (cervical, thoracic and lumbar) was considered the second most prevalent complaint, affecting approximately 13.5% of the population. It is estimated that globally 39% of the population will have at least one episode of back pain throughout their lives. In episodes of pain greater than 12 weeks (classified as chronic lower back pain), the prognosis is unfavorable and is highly associated with high treatment costs and work absenteeism.

Non-specific low back pain" [NSLBP] is defined as, low back pain that is not attributable to a recognizable or known specific pathology - bone disorder in the spine [fracture], radicular nerve compression, slipped intervertebral disk, stenosis in lumbar spine, inflammatory disorder of spine [ankylosing spondylitis], cauda equine syndrome, congenital back disorder, infection in the spine [discitis], tumour in lumbar area, osteoporosis, meningitis, Cancer, HIV, autoimmune disorder [RA].

DETAILED DESCRIPTION:
HYPOTHESIS:

Null hypothesis: There is significant effects of dry needling with conventional physiotherapy treatment as compared to Kinesio Taping with conventional physiotherapy treatment.

Alternate hypothesis: There is no significant effects of dry needling with conventional physiotherapy treatment as compared to Kinesio Taping with conventional physiotherapy treatment.

OBJECTIVES:

The aim of this study is:

* To determine the effects of dry needling in management of mechanical low back pain.
* To determine the effects of kinesio taping in management of mechanical low back pain.
* To determine the quality of life in patient with mechanical low back pain.
* To determine the varying degree of disability measure in patient with mechanical low back pain.

MATERIAL AND METHODS

3.1. Study Design Study will be a randomized control trial (RCT).

3.2. Settings The study will be conducted in the Rawal General and Dental Hospital Islamabad and Al-Nafees hospital Islamabad.

3.3. Duration of Study The duration of study will be completed in 04 months after approval of synopsis.

3.4. Sample Size Thirty patients will be enrolled in the study. Patients will be divided into groups i.e; 15 patients in each group

3.5. Sampling Technique Non probability convenient sampling. 3.6. Assessment: A pre-intervention assessment will be performed to each participant before they will be randomly assigned to kinesio taping group or dry needling group with physical therapy intervention and outcome measures will be recorded before the intervention i.e; baseline assessment ,after 2 weeks of intervention and after four weeks of treatment. After treatment, patients will be performed post-intervention assessment.

3.7. INTERVENTION: Participants will be divided into two groups Group 1: control group in which kinesiotaping with conventional physical therapy treatment (modalities including transcutaneous electrical nerve stimulation (TENS); electrical muscle stimulation (EMS); and interferential current (IFC). Physical agents including ultrasound, hot packs, and cold packs. Exercise including McKenzie exercises) will be administered.

Group 2: experimental group in which dry needling with conventional physical therapy treatment modalities including transcutaneous electrical nerve stimulation (TENS); electrical muscle stimulation (EMS); and interferential current (IFC). Physical agents including ultrasound, hot packs, and cold packs. Exercise including McKenzie exercises) will be administered.

3.8. Treatment plan: There will be a 4 weeks treatment plan consisting of 12 sessions. On each week 3 sessions will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Patient with age of 18 and above with non-specific chronic low back pain.
* Back pain of mechanical origin, apparently without a defined cause, for at least 12 weeks duration.
* Participants had not had any physical therapy treatment in the past six months and had never used Kinesio Taping and dry needling technique.
* Being asymptomatic, latent MTrPs in the muscle of lumbar region (pain during examination).
* The absence of skin allergies, Palpable taut bands (if muscle accessible).
* Recognition of usual local pain suffered by the patient pressing on the sensitive nodule on the taut bands (focally). (identification of active MTPs).
* Painful restriction of the full range of motion on passive stretching.
* The consent to physical examination, dry needling and kinesio taping application.

Exclusion Criteria:

* • Severe injury in the last 12 months.

  * Previous spinal surgical intervention, neurological diseases or musculoskeletal dis-orders, pharmacological treatment at present.
  * infection, open wound, rash, decreased blood circulation in the treatment area
  * A pacemaker, or epilepsy, presence of skin diseases and pregnancy
  * Serious spinal pathologies such as a tumor, an inflammatory disease or former fracture of L1-S1, symptoms of spinal stenosis, disc protrusion or nerve root compromise and degeneration established in more than two levels
  * Subjects who had used or had prior knowledge of the Kinesio Taping and dry needling method.
  * generalized chronic pain, fibromyalgia, clinical sign of radiculopathy and peripheral nervous system diseases
  * spondylolysis with or without spondylolisthesis, arthritis or osteoporosis and Congenital or acquired deformity
  * ongoing psychiatric or somatic disease that excluded either one or both treatment alternatives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
comparison of dry needling and kinesio taping in management of mechanical low back pain. | 6 months
  mechanical low back pain will be measured using Roland Morris low back questionnaire and Pain Numeric Rating scale calculated as mean score.

SECONDARY OUTCOMES:
Quality of life in patient with mechanical low back pain | 6 months
  Determine the quality of life in patient with mechanical low back pain by using WHO-QOL Questionnaire in term of domain score.

CONTACTS AND LOCATIONS:
Overall Officials: Adeela Asad, m.phil, Principal Investigator — Rawal Institue of Health Sciences Islamabad
Locations (1):
- Adeela Asad, Islamabad, Federal Capital, Pakistan